CLINICAL TRIAL: NCT01307566
Title: Evolution With CPAP Treatment of a Cohort of Type 2 Diabetic Patients With Moderate to Severe Apnea-hypopnea Syndrome and Poor Glycemic Control
Brief Title: Evolution With CPAP Treatment of a Cohort of Type 2 Diabetic Patients With Apnea-hypopnea Syndrome
Acronym: DM2-CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Granollers (Other)
Collaborators: EsteveTeijin Healthcare (Other)
Responsible Party: Principal Investigator, marta torrella, Chest Physician in Unitat de Pneumologia, Hospital de Granollers
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM2-CPAP
Record Dates: First submitted 2011-02-11; First posted 2011-03-03 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Sleep Apnea; Type 2 Diabetes
MeSH Terms: conditions — Sleep Apnea Syndromes; Diabetes Mellitus, Type 2 | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Continuous Positive Airway Pressure (Experimental): Continuous Positive Airway Pressure (CPAP)
  Interventions: Device: Continuous Positive Airway Pressure CPAP

INTERVENTIONS:
Device: Continuous Positive Airway Pressure CPAP — CPAP treatment
  Other Names: no other name

SUMMARY:
The main purpose of this study is to measure the evolution of hemoglobin A1c level after treatment with CPAP in a cohort of type 2 diabetes mellitus patients with poor glycemic control and associated moderate or severe obstructive sleep apnea.

DETAILED DESCRIPTION:
Subjects with poorly controlled type 2 diabetes are a high cardiovascular risk group in which a high prevalence of moderate to severe sleep apnea is expected. Studies based on interstitial glycemic measurement demonstrate a reduction in glucose levels when treating sleep apnea with CPAP. Nevertheless, the effectiveness of CPAP in improving glycemic control has been questioned as most studies have failed to demonstrate a reduction in hemoglobin A1c (HbA1C) level over time. Most of these studies have limitations such as a short follow-up or a suboptimal fulfillment of CPAP treatment. We hypothesize that treating moderate to severe sleep apnea with CPAP will improve glycemic control (measured by HbA1C) at 14 weeks in good compliers and that this improvement will be sustained at one year. We aim to test this hypothesis in consecutive type 2 diabetes patients on stable treatment with HbA1c ≥7% in routine outpatient visits in our Diabetes, Nutrition and Endocrinology Unit. After providing informed consent, patients will be screened for sleep apnea by nocturnal oximetry followed by a diagnostic respiratory polygraphy. Those patients with obstructive sleep apnea with an apnea-hypopnea index ≥20 will be invited to enter the study. After a 3-month observation period without any intervention to rule out a potential influence of entering the study on HbA1C levels, patients will be treated with CPAP. HbA1C levels will be measured at baseline, after 14 weeks, and thereafter every 14 weeks until completing one year of treatment. Other endocrine, metabolic and cardiovascular risk variables will be determined at baseline and at 14 weeks of the intervention.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes on stable treatment for the last three months and HbA1C ≥ 7%
* Obstructive Sleep Apnea with and apnea-hypopnea index ≥20
* Acceptance of a therapeutic trial with CPAP

Exclusion criteria:

* Race: non caucasic
* Blood level of hemoglobin <10 in women or <11 in men or iron defitiency or hemoglobinopathy
* Glomerular filtration rate < 30
* Habitual sleeping time <6 hours per night
* Nocturnal work, shift work or unsual sleeping schedule
* Primary severe insomnia or secondary to restless legs syndrome
* Major or non stable psychiatric disorder
* Treatment with corticosteroids
* Chronic respiratory disorders that may require corticosteroids or cause respiratory insufficiency or FEV1/FVC<0.7 with FEV1<50 in spirometry
* Predominant nocturnal hypoventilation pattern
* Cardiac failure
* Alcohol abuse
* Active CPAP treatment
* Previous surgery for sleep apnea
* Severe nasal obstruction
* Illiteracy

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobine A1C from baseline | 14, 28, 42 and 56 weeks after initial intervention.

SECONDARY OUTCOMES:
Blood levels of fasting glucose from baseline | 14 weeks after initial intervention
Self measured capillary glucose profile | 14 weeks after initial intervention
Evening saliva collection for cortisol assay | 14 weeks after initial intervention
Noninvasive 24-hour ambulatory blood pressure monitoring | 14 weeks after initial intervention.
Analysis of urine to assess albumin to creatinine ratio | 0, 14, 28, and 56 weeks after initial intervention.
Blood levels of fasting insulin | 14 weeks after initial intervention
Blood levels of total cholesterol | 14 weeks after initial intervention
Blood levels of cholesterol HDL | 14 weeks after initial intervention
Blood levels of tryglicerids | 14 weeks after initial intervention
International Physical Activity Questionnaire | 14 weeks after initial intervention
Epworth Sleepiness Scale | 14 weeks after initial intervention
SF-36 v2 Health Survey | 14 weeks after initial intervention
subjective quantity and quality of sleep reported in a sleep log | 14 weeks after initial intervention
Change in ratio albumine to creatinine from baseline | 14, 28, 42 and 56 weeks after initial intervention

CONTACTS AND LOCATIONS:
Overall Officials: Marta Torrella, M.D., Principal Investigator — Granollers General Hospital
Locations (1):
- Granollers General Hospital, Granollers, Barcelnoa, Spain